CLINICAL TRIAL: NCT07036146
Title: Single-center Transversal Observational Study on the Evaluation of S100B Changes in Subjects Attending the Emergency Department With Head Trauma
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Locatelli, Medical doctor, IRCCS San Raffaele
Other Study IDs: SMART
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Head Trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venus blood withdrawal (approximately 3-5 mL)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects admitted at the ED with head trauma, regardless of age or gender

SUMMARY:
The aim of the study is to evaluate blood levels of the calcium-binding protein S100B as a diagnostic biomarker for the management of patients with suspected traumatic brain injury. With a sensitivity of 97% and a negative predictive value greater than 99%, S100B measurement can predict the absence of brain injury, supporting risk stratification and the safe discharge of low-risk patients. This, in turn, may reduce the need for imaging studies and shorten emergency department stays. The management of patients enrolled in the study will be identical to that of non-enrolled patients. The only difference is that patients in the study will undergo a blood draw, whereas in routine practice blood tests are not mandatory (although they are often performed).

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of death and hospital admissions worldwide, with over 50 million new cases occurring globally annually. Based on the severity, brain traumas have been classified in four different categories: Minimal, Mild, Moderate and Severe TBI. Mild and Moderate TBI (mTBI), represents the vast majority of TBIs occurring in the ED. Imaging techniques, such as computed tomography (CT), are traditionally the most widely used diagnostic method in evaluating a patient with suspected mTBI. However, only approximately 16% of patients attending the ED with suspected mTBI present intracranial lesions (proved with imaging techniques). Furthermore, the diagnostic process based on imaging techniques involves an average stay in the ED of approximately 7 hours. Despite the low diagnostic yield, the high cost and the potential side effect of the ionizing radiation, the use of imaging techniques is supported on the basis that even a mTBI can hide a serious, life-threatening injury.

In this context, the beta subunit of the calcium binding protein S100B has emerged as a highly diagnostic biomarker in the management of TBI, and in particular for mTBI, if the measurement is performed within the first hours of trauma. S100B can be detected with a simple and rapid routine venous blood test, making its use minimally invasive for the patient and extremely more efficient (both in terms of costs and time) for the hospital. Thanks to a sensitivity of 97% associated with a negative predictive value >99%, the S100B dosage can predict the absence of brain damage, facilitating risk stratification and safe discharge of low-risk patients allowing the reduction of the number of imaging tests, and consequently the patient's length of stay in the ED.

The S100B dosage is therefore an objective tool for patient triage. It is simpler and faster to perform than imaging techniques and involves reduced treatment costs which can be estimated at approximately 100 euros per patient.

The implementation of the S100B dosage in a clinical/diagnostic routine becomes even more important in pediatric settings. It has been shown that exposure to ionizing radiation at a young age (0-19 years) can increase the risk of cancer by up to 24%. In this context, S100B has proven to be a very promising biomarker for children with mTBI. A meta-analysis of eight studies highlighted for S100B a sensitivity and a negative predictive value, for intracranial lesions, both of 100%. Implementation of a modified PECARN (Pediatric Emergency Care Applied Research Network) rule, which includes measurement of S100B protein, reduced by 70% the number of diagnostic imaging investigations needed to identify mTBI in a pediatric population.

Recently the Scandinavian Neurotrauma Committee (SNC) recommended serum S100B dosing as a biomarker for low-risk mild traumatic brain injury. Based on this evidence and considerations, we believe it is of primary importance to carry out a study aimed at the future implementation, also in our hospital, of the S100B dosage.

The study mainly aims at:

1. registering the fluctuations in the quantification of the S100B protein in cases of mTBI
2. characterizing the sensitivity and the negative predictive value of the test for an efficient stratification of the prognosis of different entities of head trauma

The dosage of S100B at the OSR will be carried out via the COBAS8000 (Roche) large automation line, already present in OSR. The reagents are commercially available. This will allow to obtain results in a very short time (within minutes) and at very low costs.

Secondly, the study aims to store the biological samples (serum) at the OSR Biological Resources Center. The samples will be used later to evaluate the diagnostic potential of novel blood markers of brain damage that have recently emerged in the literature and could, in the future, be part together with S100B of a highly sensitive analytical panel. These biomarkers are; the glial fibrillary acidic protein (G-FAP), the ubiquitin c-terminal hydrolase L1 (UCH-L1) and the neurofilament light (NfL).

As for S100B, the dosage of G-FAP, UCH-L1 and NfL will be carried out at OSR, using the COBAS8000 large automation line (Roche).

ELIGIBILITY:
Inclusion Criteria:

* Either males or female patients, aged 0-100 years, who signed the study informed consent, including pregnant and breastfeeding women admitted at the ED with a head trauma occurred less than 6 hour prior to admission to the ED. Unconscious patients will still be enrolled if they regain consciousness within 6 hours of the trauma

Exclusion Criteria:

* unconscious patients as well as patients for whom the head trauma occurred at least 6 hours before presenting to the emergency room

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Either males or female patients, aged 0-100 years, who signed the study informed consent, including pregnant and breastfeeding women admitted at the ED with a head trauma occurred less than 6 hour prior to admission to the ED.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Verify and confirm the correlation between blood S100B levels (>0.1 µg/L) and head trauma severity as determined by the GCS and clinical symptoms | Blood sampling at day 0 (at ED admission)
  The concentration of S100B in the blood will be measured in patients admitted to the Emergency Department with head trauma. Correlations between blood S100B levels and head trauma severity as determined by the GCS and clinical symptoms will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed at the IRCCS San Raffaele Hospital with no need to share individual participant data